CLINICAL TRIAL: NCT05410470
Title: Efficacy and Safety of Ruxolitinib in Patients With Myelofibrosis: A Retrospective Multicenter Study
Brief Title: Efficacy and Safety of Ruxolitinib in Patients With Myelofibrosis
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: QiluH MF
Record Dates: First submitted 2022-05-23; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MF patients who received ruxolitinib treatment
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib

SUMMARY:
Ruxolitinib is a Janus kinase (JAK) 1/2 inhibitor currently used in the treatment of Myelofibrosis (MF). Ruxolitinib confirmed improvements in splenomegaly, MF-related symptoms and survival benefit in COMFORT and JUMP studies. At present, the real-world data on the efficacy and safety of ruxolitinib in the treatment of MF in China is still insufficient. The aim of this study was to evaluate the efficacy and safety of ruxolitinib in patients with MF and to provide guidance for the usage of ruxolitinib in MF in China.This was a retrospective, multicenter study of MF patients who received ruxolitinib treatment in Shandong province from August 2012 to December 2021. Data were analyzed using SPSS. Overall survival (OS) and Event-free survival (EFS) were estimated using the Kaplan- Meier method.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years with a diagnosis of primary or secondary MF by World Health Organization and International Working Group for Myeloproliferative Neoplasms Research and Treat- ment (IWG-MRT) criteria;
2. Received ruxolitinib treatment for ≥3 months.

Exclusion Criteria:

1. Malignant tumors with other progression or myelofibrosis secondary to other diseases;
2. Exclude myelofibrosis patients after splenectomy;
3. Patients with poor compliance with case follow-up or lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MF patients including primary and secondary MF patients who received ruxolitinib treatment are going to be recruited.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a ≥35% reduction in palpable spleen volume from baseline. | From Week 0 through Week 24
  Reduction in spleen volume is measured by magnetic resonance imaging/computerized tomography (MRI/CT).

SECONDARY OUTCOMES:
The proportion of patients with ≥50% reduction in Total Symptom Score (TSS) from baseline. | From Week 0 through Week 24
  TSS is assessed by the MPN-10.